CLINICAL TRIAL: NCT04574843
Title: Middle Meningeal Artery Embolization With Liquid Embolic Agent for Treatment of Chronic Subdural Hematoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Humain Baharvahdat, Associate Professor, Mashhad University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 990631
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Chronic Subdural Hematoma
Keywords: chronic subdural hematoma; embolization; middle meningeal artery; liquid embolic agent
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — ethylene-vinyl alcohol copolymer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embolization arm (Experimental): Intervention: Embolization of middle meningeal artery Device: Onyx, squid, Phil
  Interventions: Procedure: Embolization of MMA

INTERVENTIONS:
Procedure: Embolization of MMA — embolization of MMA with one of following liquid embolic agents (Onyx-Squid-Phil)
  Other Names: Onyx; Squid; Phil

SUMMARY:
The study evaluates the clinical and imaging outcome of middle meningeal artery (MMA) embolization with liquid embolic agent for treatment of chronic subdural hematoma (CSDH)

DETAILED DESCRIPTION:
This study is a prospective one arm trial designed to assess the safety and efficacy of MMA embolization with liquid embolic agents (onyx/squid/Phil) as the main treatment of CSDH.

The subjects are enrolled in the study according to inclusion and exclusion criteria. Imaging and clinical presentations of patients are recorded. Within 48 hours of embolization, patients are assessed with clinical examination and with a brain CT scan to evaluate in any change in their symptoms and CSDH volume. 2-4 weeks after embolization, patients are evaluated in clinic for any change in their symptoms and signs. 60 days after embolization patients are examined clinically and are assessed for SDH volume change in CT scan and MRI.

If there is any significant increase in CSDH volume or any deterioration of patient, evacuation of hematoma is considered.

MMA embolization is performed under general anesthesia using biplane or monoplane angiography. Femoral or radial accesses are used. Guiding catheter is advanced into external carotid artery in corresponding side. The corresponding MMA is catheterized distally by micro-catheter and is embolized by liquid embolic agents. Patients are discharge next day if they are stable.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed chronic or subacute subdural hematoma
2. Patients had symptoms/signs associated with chronic or subacute subdural hematoma: severe headache, hemiparesis/monoparesis, dementia, aphasia/dysphasia, loss of consciousness, ...
3. Asymptomatic large chronic/subacute hematoma after 6-8 weeks of failed conservative treatment

Exclusion Criteria:

1. presentation with coma (GCS =< 8)
2. patients needs emergent evacuation of hematoma,
3. patients could not participate in 60 days follow-up
4. pregnant patients
5. acute subdural hematoma
6. contraindication to contrast
7. contradiction to angiography
8. difficult access to MMA due to anatomical variation
9. contraindication to liquid embolic agent
10. unmanaged/uncontrollable bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of CSDH regression | 60 dyas
  Volume reduction of CSDH in follow-up imaging (CT/MRI) 60 days after embolization

SECONDARY OUTCOMES:
Incidence of CSDH progression or recurrence | 60 days
  Increase in volume of CSDH
Incidence of new neurological deficit (ND) | 60 days
  ND includes: dementia, memory loss, cognitive problems, monoparesis/hemiparesis, cranial nerve paresis, dysphasia/aphasia
incidence of Death | 60 days
Incidence of new ischemic stroke | 60 days
  new ischemia in imaging (DWI/MRI or CT scan) within 60 days of operation
Incidence of myocardial infarction/myocardial ischemia | 60 days
  new ischemic heart attack within 60 days of operation
Incidence of embolization complication in brain | 48 hours
  cranial nerve palsy (especially VII), vision loss (ophthalmic/retinal artery occlusion), ...
incidence of embolization complication out of brain | 15 days
  puncture hematoma, major artery dissection, new renal failure, ...

CONTACTS AND LOCATIONS:
Overall Officials: Humain Baharvahdat, MD, Study Director — Department of Neurosurgery, Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Ghaem Hospital, Mashhad University of Medical Sciences, Mashhad, Iran

IPD SHARING:
Plan to Share IPD: No